CLINICAL TRIAL: NCT04036656
Title: Single-center, Randomized, Double-blind, Placebo-controlled, Single Dose Ascending Trial of SYHA 136 Tablets in Healthy Subjects
Brief Title: Phase I Study of Direct Coagulation Factor Xa Inhibitor SYHA136 Tablets in Chinese Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SYHA136201901/PRO-I
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1:SYHA136 0.5 mg or Placebo matching SYHA136 0.5 mg (Experimental): Participants will receive a single oral dose of SYHA136 0.5 mg or Placebo matching SYHA136 0.5 mg under fasted conditions.
  Interventions: Drug: SYHA136 0.5 mg; Drug: Placebo matching SYHA136 0.5 mg
- Cohort 2:SYHA136 1 mg or Placebo matching SYHA136 1 mg (Experimental): Participants will receive a single oral dose of SYHA136 1 mg or Placebo matching SYHA136 1 mg under fasted conditions.
  Interventions: Drug: SYHA136 1 mg; Drug: Placebo matching SYHA136 1 mg
- Cohort 3:SYHA136 2.5 mg or Placebo matching SYHA136 2.5 mg (Experimental): Participants will receive a single oral dose of SYHA136 2.5 mg or Placebo matching SYHA136 2.5 mg under fasted conditions.
  Interventions: Drug: SYHA136 2.5 mg; Drug: Placebo matching SYHA136 2.5 mg
- Cohort 4:SYHA136 5 mg or Placebo matching SYHA136 5 mg (Experimental): Participants will receive a single oral dose of SYHA136 5 mg or Placebo matching SYHA136 5 mg under fasted conditions.
  Interventions: Drug: SYHA136 5 mg; Drug: Placebo matching SYHA136 5 mg
- Cohort 5:SYHA136 10 mg or Placebo matching SYHA136 10 mg (Experimental): Participants will receive a single oral dose of SYHA136 10 mg or Placebo matching SYHA136 10 mg under fasted conditions.
  Interventions: Drug: SYHA136 10 mg; Drug: Placebo matching SYHA136 10 mg
- Cohort 6:SYHA136 20 mg or Placebo matching SYHA136 20 mg (Experimental): Participants will receive a single oral dose of SYHA136 20 mg or Placebo matching SYHA136 20 mg under fasted conditions.
  Interventions: Drug: SYHA136 20 mg; Drug: Placebo matching SYHA136 20 mg
- Cohort 7:SYHA136 35 mg or Placebo matching SYHA136 35 mg (Experimental): Participants will receive a single oral dose of SYHA136 35 mg or Placebo matching SYHA136 35 mg under fasted conditions.
  Interventions: Drug: SYHA136 35 mg; Drug: Placebo matching SYHA136 35 mg
- Cohort 1:SYHA136 50 mg or Placebo matching SYHA136 50 mg (Experimental): Participants will receive a single oral dose of SYHA136 50 mg or Placebo matching SYHA136 50 mg under fasted conditions.
  Interventions: Drug: SYHA136 50 mg; Drug: Placebo matching SYHA136 50 mg

INTERVENTIONS:
Drug: SYHA136 0.5 mg — oral tablet
  Arms: Cohort 1:SYHA136 0.5 mg or Placebo matching SYHA136 0.5 mg
Drug: SYHA136 1 mg — oral tablet
  Arms: Cohort 2:SYHA136 1 mg or Placebo matching SYHA136 1 mg
Drug: SYHA136 2.5 mg — oral tablet
  Arms: Cohort 3:SYHA136 2.5 mg or Placebo matching SYHA136 2.5 mg
Drug: SYHA136 5 mg — oral tablet
  Arms: Cohort 4:SYHA136 5 mg or Placebo matching SYHA136 5 mg
Drug: SYHA136 10 mg — oral tablet
  Arms: Cohort 5:SYHA136 10 mg or Placebo matching SYHA136 10 mg
Drug: SYHA136 20 mg — oral tablet
  Arms: Cohort 6:SYHA136 20 mg or Placebo matching SYHA136 20 mg
Drug: SYHA136 35 mg — oral tablet
  Arms: Cohort 7:SYHA136 35 mg or Placebo matching SYHA136 35 mg
Drug: SYHA136 50 mg — oral tablet
  Arms: Cohort 1:SYHA136 50 mg or Placebo matching SYHA136 50 mg
Drug: Placebo matching SYHA136 0.5 mg — oral tablet
  Arms: Cohort 1:SYHA136 0.5 mg or Placebo matching SYHA136 0.5 mg
Drug: Placebo matching SYHA136 1 mg — oral tablet
  Arms: Cohort 2:SYHA136 1 mg or Placebo matching SYHA136 1 mg
Drug: Placebo matching SYHA136 2.5 mg — oral tablet
  Arms: Cohort 3:SYHA136 2.5 mg or Placebo matching SYHA136 2.5 mg
Drug: Placebo matching SYHA136 5 mg — oral tablet
  Arms: Cohort 4:SYHA136 5 mg or Placebo matching SYHA136 5 mg
Drug: Placebo matching SYHA136 10 mg — oral tablet
  Arms: Cohort 5:SYHA136 10 mg or Placebo matching SYHA136 10 mg
Drug: Placebo matching SYHA136 20 mg — oral tablet
  Arms: Cohort 6:SYHA136 20 mg or Placebo matching SYHA136 20 mg
Drug: Placebo matching SYHA136 35 mg — oral tablet
  Arms: Cohort 7:SYHA136 35 mg or Placebo matching SYHA136 35 mg
Drug: Placebo matching SYHA136 50 mg — oral tablet
  Arms: Cohort 1:SYHA136 50 mg or Placebo matching SYHA136 50 mg

SUMMARY:
The trial used single-center, randomized, double-blind, placebo-controlled, single-dose ascending study.

The trial planned to enroll fifty-six healthy volunteers. The subjects were allocated to eight dose groups, including 0.5 mg (3+1), 1 mg (3+1), 2.5 mg (6+2), 5 mg (6+2), 10 mg (6+2), 20 mg (6+2), 35 mg(6+2) and 50 mg (6+2). Each dose group was allocated test drugs and placebos according to the proportion of subjects in the brackets mentioned above.

ELIGIBILITY:
Inclusion Criteria:

1. When subject signs the informed contest, 18≤ age ≤ 40, Male or female;
2. Body weight: male ≥50 kg, female ≥45 kg. Body mass index (BMI) of 19.0 to 26.0 kg/m², inclusive;
3. Subject's with normal or or abnormity without clinical significance judged by the investigator by physical examination, vital signs, electrocardiogram, blood routine, blood biochemistry, coagulation tests, fecal occult blood, urine routine, serological tests and other important indicators;
4. All subjects who adopt effective non-hormonal contraceptive measures (such as condoms, intrauterine devices without drugs, etc.) from the signing of informed consent to three months after the end of the study;
5. Subjects who voluntarily signed the informed consent and are able to cooperate to complete the test according to the protocal.

Exclusion Criteria:

1. Allergic history to more than one drug or other serious allergic rhistory;
2. Serious diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders or other diseases (such as history of psychosis, malignant tumors, etc.)In the past or now, which were not suitable for clinical trials.
3. History of abnormal bleeding or coagulation disorders (e.g. prone to bruising, gum bleeding, prolonged bleeding after tooth extraction, joint hemorrhage, menorrhagia, postpartum hemorrhage, vitamin K deficiency, haemorrhagic diseases caused by acquired coagulation factor antibodies, trauma, wound or post-operative bleeding, etc.);
4. History of severe head trauma in 2 years;
5. Severe gastrointestinal diseases occurred within three months before signing informed consent, which affected drug absorption;
6. Have a disease which Haemorrhage could cause serious consequences, such as peptic ulcer;
7. Had undergone surgery within six months before signing the informed consent; planned to undergo surgery (including cosmetic surgery, dental surgery and oral surgery) within two weeks after the end of the trial; or planned to take part in vigorous exercise (including physical contact exercise or collision exercise) during the trial;
8. Bleed or donated more than 400 mL within three months before signing informed consent, or planned to donate blood during the study or within one month after the end of the trial;
9. Have taken any prescription drugs, nonpreserip drugs, biological products, traditional Chinese medicines, herbal medicines, vitamin dietary supplements and health products within four weeks before signing the informed consent or use oral long-acting contraceptives or implanted long-acting contraceptives;
10. Subjects participating in other clinical trials and taking trial products, or participated in any other clinical trials of drugs within three months before signing the informed consent;
11. History of drugs or drug abuse or alcoholics or drug abuse screening shows positive response;
12. current or past alcoholics (drinking more than 14 standard units per week, 1 Standard unit containing 14g alcohol, such as 360 mL beer or 40% spirits or 150 mL wines with 45 mL alcohol), or alcohol breath test positive;
13. Smokers: The average daily smoking volume was more than 5 cigarettes within six months before signing the informed consent;
14. Habitually consume excessive caffeine-containing beverages or foods, or foods that may affect drug metabolism within four weeks before signing informed consent. Such as: coffee (no more than 1100 mL per day), tea (no more than 2200 mL per day), cola (no more than 2200 mL per day), functional drinks (no more than 1100 mL per day), chocolate (no more than 510 g per day);
15. Positive with serum immunological test for HBsAg, Anti-HCV, Anti-HIV or Anti-TP;
16. QTc interval≥450 ms, electrocardiogram abnormality with clinical significance, or prolonged history of QTc interval;
17. Abnormal results of chest X-ray (posterior and anterior) with clinical significance;
18. Female subjects: positive pregnancy tests or pregnant or breast-feeding or planning to conceive, who plan to conceive within three months from the signing of informed consent to the end of the study; male subjects: whose partners plan to conceive or plan to donate sperm within three months from the signing of informed consent to the end of the study;
19. Not suitable for this trial according to the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From Screening period to 12 Days Post dose
  Number of participants that experience Adverse Events (AEs)
Serious Adverse Events (SAEs) | From Screening period to 12 Days Post dose
  Number of participants that experience Serious Adverse Events (SAEs)
clinically significant laboratory assessment abnormalities | Up to 72 hours Post dose
  Number of participants with clinically significant laboratory assessment abnormalities
clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to 72 hours Post dose
  Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities
clinically significant physical examination abnormalities | Up to 72 hours Post dose
  Number of participants with clinically significant physical examination abnormalities

SECONDARY OUTCOMES:
Area Under the concentration-time curve from time zero to time of the Last Measurable Concentration (AUC0-tlast) | Up to 72 hours Post dose
  PK Assessment - Area Under the concentration-time curve from time zero to time of the Last Measurable Concentration (AUC0-tlast)
Area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to 72 hours Post dose
  PK Assessment - Area under the concentration-time curve from time 0 to infinity (AUCinf)
Maximum observed concentration (Cmax) | Up to 72 hours Post dose
  PK Assessment - Maximum observed concentration (Cmax)
Time to reach maximum observed concentration (Tmax) | Up to 72 hours Post dose
  PK Assessment - Time to reach maximum observed concentration (Tmax)
Terminal elimination half-life (t1/2) | Up to 72 hours Post dose
  PK Assessment - Terminal elimination half-life (t1/2)
Apparent total body clearance (CL/F) | Up to 72 hours Post dose
  PK Assessment - Apparent total body clearance (CL/F)
Apparent volume of distribution (Vz/F) | Up to 72 hours Post dose
  PK Assessment - Apparent volume of distribution (Vz/F)
Amount of SYHA136 excreted in urine (Aeu) | Up to 72 hours Post dose
  PK Assessment - Amount of SYHA136 excreted in urine (Aeu)
Renal clearance (CLr) | Up to 72 hours Post dose
  PK Assessment - Renal clearance (CLr)
Activated Partial Thromboplastin Time(aPTT) | Up to 48 hours Post dose
  PD Assessment-Activated Partial Thromboplastin Time(aPTT)
Fibrinogen(Fbg) | Up to 48 hours Post dose
  PD Assessment-Fibrinogen(Fbg)
Thrombin Time(TT) | Up to 48 hours Post dose
  PD Assessment-Thrombin Time(TT)
International Normalized Ratio(INR) | Up to 48 hours Post dose
  PD Assessment-International Normalized Ratio(INR)
Anti-coagulation Factor Xa assays(AXA) | Up to 48 hours Post dose
  PD Assessment-Anti-coagulation Factor Xa assays(AXA)

IPD SHARING:
Plan to Share IPD: No